CLINICAL TRIAL: NCT01413516
Title: A Two-Part Pilot Study of Dosing, Safety and Efficacy of Varenicline Initiated During an Acute Smoke-free Hospitalization and Continued Post-Hospitalization
Brief Title: Varenicline In-Patient Study
Acronym: VIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Judith Prochaska, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIP
Record Dates: First submitted 2011-08-03; First posted 2011-08-10 (Estimated); Results first posted 2016-12-30 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Smoking Cessation
Keywords: Varenicline; Placebo; Inpatient
MeSH Terms: conditions — Smoking Cessation | interventions — Sugars; Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Control (Placebo Comparator): Smoking cessation counseling with placebo comparator
  Interventions: Behavioral: Smoking cessation counseling; Drug: Placebo
- Experimental: Varenicline (Active Comparator): Smoking cessation counseling with varenicline
  Interventions: Behavioral: Smoking cessation counseling; Drug: Varenicline

INTERVENTIONS:
Behavioral: Smoking cessation counseling — Counseling sessions provided by a trained smoking counselor
Drug: Placebo — Sugar pill without any active medication
  Other Names: sugar pill (control)
  Arms: Placebo Control
Drug: Varenicline — Varenicline (an approved medication for smoking cessation)
  Other Names: Chantix
  Arms: Experimental: Varenicline

SUMMARY:
This Investigator Initiated Research Award (IIR Award #WS981308) is a two-part pilot study that aims to examine acceptability and feasibility of varenicline use during an acute (72-hr) smoke-free hospitalization (Part 1) and 4-weeks post-hospitalization (Part 2).

DETAILED DESCRIPTION:
The sample will be hospitalized patients smoking at least 10 cigarettes/day prior to hospitalization. Intention to quit smoking will not be required for study participation. Using a double-blinded, placebo-controlled, randomized design, participants will receive varenicline (0.5 mg BID as tolerated) or placebo during their hospitalization (Part 1) and will continue their study medication (placebo or active drug) for 4 weeks post-hospitalization (Part 2). Abstinence status will be examined at 4 weeks post-hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* The sample, 40 women and 40 men, will be hospitalized patients recruited from Stanford Hospital and Clinics who report smoking at least 10 cigarettes per day prior to hospitalization, have confirmed tobacco use by cotinine testing, and an expected hospitalization of at least 3 days duration from the date of study enrollment. Intention to quit smoking will not be required for study participation.

Exclusion Criteria:

- Study exclusion criteria are: dementia or other brain injury precluding ability to participate; Alzheimer's Disease; Parkinson's Disease; Huntington's Disease; meningitis; seizure disorder of a sustained nature; delirium; brain surgery; drug and/or alcohol dependence; suicidal ideation; end-stage renal disease (i.e., on dialysis); hypertensive crisis; stroke; myocardial infarction (MI) with severe cardiac damage; pregnancy or breastfeeding; non-English speaking; complete homelessness; or currently engaged in tobacco treatment. Study staff will consult with clinical staff prior to approach for study enrollment. In cases of severe renal impairment (estimated creatinine clearance <30 mL/min), medical staff will consult with participants' physician to assess the appropriateness for study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith J Prochaska, PhD, MPH, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Sugar Pill Without Any Active Medication: Smoking counseling, Placebo: Placebo comparator
  Interventions:
  * Behavior: smoking counseling
  * Drug: placebo (sugar pill without any active medication)
  Smoking counseling: Counseling sessions provided by a trained smoking counselor during 1st day of study along with 28 day supply of placebo
  Placebo: Sugar pill without any active medication
- Experimental: Varenicline: Smoking counseling, Varenicline: Experimental
  Interventions:
  * Behavioral: smoking counseling
  * Drug: varenicline
  Smoking counseling: Counseling sessions provided by trained smoking counselor during 1st day of study along with 28 day supply of varenicline
  Varenicline: Varenicline (an approved medication for smoking cessation)
Period: Overall Study
Arm/Group | Control: Sugar Pill Without Any Active Medication | Experimental: Varenicline
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Sugar Pill Without Any Active Medication: Smoking counseling, Placebo: Placebo comparator
  Interventions:
  * Behavior: smoking counseling
  * Drug: placebo (sugar pill without any active medication)
  Smoking counseling: Counseling sessions provided by a trained smoking counselor along with placebo during 1st day of study
  Placebo: Sugar pill without any active medication
- Experimental: Varenicline: Smoking counseling, Varenicline: Experimental
  Interventions:
  * Behavioral: smoking counseling
  * Drug: varenicline
  Smoking counseling: Counseling sessions provided by trained smoking counselor along with varenicline
  Varenicline: Varenicline (an approved medication for smoking cessation)
- Total: Total of all reporting groups
Arm/Group | Control: Sugar Pill Without Any Active Medication | Experimental: Varenicline | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (14) | 48 (13) | 50 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: 7 Day Point Prevalence Abstinence From All Forms of Tobacco
Description: Self report of being quit for 7 continuous days at the time of the 4-week follow-up survey confirmed by saliva cotinine or urine anabasine verification.
Time Frame: 4 weeks after beginning study
Measure: Number; unit: participants
Groups:
- Sugar Pill Without Any Active Medication: Smoking counseling, Placebo: Placebo comparator
  Interventions:
  * Behavior: smoking counseling
  * Drug: placebo (sugar pill without any active medication)
  Smoking counseling: Counseling sessions provided by a trained smoking counselor along with placebo during 1st day of study
  Placebo: Sugar pill without any active medication
Arm/Group | Sugar Pill Without Any Active Medication | Experimental: Varenicline
Number analyzed (Participants) | 8 | 9
participants | 2 | 2

ADVERSE EVENTS:
Description: assessed by self-report at every time point
Arm/Group | Control: Sugar Pill Without Any Active Medication | Experimental: Varenicline
Serious Adverse Events (participants affected / at risk) | 0/8 | 2/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control: Sugar Pill Without Any Active Medication (N=8) | Experimental: Varenicline (N=9)
Leg amputation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — This was a planned re-hospitalization for a follow-up surgical procedure. Participant reported finishing his 4-week course of study medication on the day prior to re-hospitalization.
Renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1) — This adverse event occurred after the participant was scheduled to finish the 4 week course of of study medication. Participant was unable to recall whether taking study medication when the onset of the events described in the narrative occurred.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No